CLINICAL TRIAL: NCT03059212
Title: rTMS in Facilitation of Working Memory in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, principal investigator, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-10-018A
Record Dates: First submitted 2017-01-16; First posted 2017-02-23 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease
Keywords: working memory; parkinson's disease; cognition; rTMS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Real rTMS, sham rTMS
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High frequency rTMS (Experimental): Real rTMS, one session per day, for 10 days
  Interventions: Device: rTMS
- High frequency rTMS with cognitive training (Experimental): Real rTMS and cognitive training, one session per day, for 10 days
  Interventions: Device: rTMS; Behavioral: Cognitive training program
- Sham rTMS (Sham Comparator): Sham rTMS, one session per day, for 10 days
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — High frequency rTMS for 3 to 10 min to increase the excitability of cortex.
Behavioral: Cognitive training program — A rehabilitation protocol that facilitates attention, memory, execution.
  Arms: High frequency rTMS with cognitive training

SUMMARY:
Ten sessions of repetitive transcranial magnetic stimulation yield ability to upregulate the function of primary motor cortex and prefrontal cortex that play key roles in motor and frontal memory processing.

DETAILED DESCRIPTION:
Excitatory (>3Hz) rTMS could facilitate the brain cortex and neuroplasticity that benefits motor control and working memory when the coil is applied over primary motor cortex or dorsolateral prefrontal cortex.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease
* With symptoms of cognitive impairments, such as memory, attention, or language decline.

Exclusion Criteria:

* History of seizure attack
* Alzheimer's disease
* With cardiac pacemaker implantation

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change of Repeatable Battery for the Assessment of Neuropsychological Status | up to 12 weeks
  This battery measures the cognitive functions including attention, memory, language, visuospatial domains.

SECONDARY OUTCOMES:
Change of Montreal Cognitive Assessment ; MoCA | up to 12 weeks
  Assessing cognitive function including delaying recall, attention, executive function, language...

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yi Tsai, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veteran General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Preston G, Anderson E, Silva C, Goldberg T, Wassermann EM. Effects of 10 Hz rTMS on the neural efficiency of working memory. J Cogn Neurosci. 2010 Mar;22(3):447-56. doi: 10.1162/jocn.2009.21209. PMID 19309294
- See also: Description Related Info — http://www.ncbi.nlm.nih.gov/pubmed/23194830
- See also: Description Related Info — http://www.ncbi.nlm.nih.gov/pubmed/21980359
- See also: Description Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19309294